CLINICAL TRIAL: NCT01615627
Title: Hypotonic Treprostinil Subcutaneous Infusion for Control of Treprostinil Related Site Pain
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No enrollment
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Dr David Langleben, Chair, Cardiology Department, Jewish General Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JGH-12-058
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Subcutaneous Treprostinil
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypotonic Treprostinil Solution (Experimental): Hypotonic Treprostinil Solution
  Interventions: Drug: HypotonicTreprostinil Solution
- Eutonic Treprostinil Solution (Active Comparator): Eutonic Treprostinil Solution
  Interventions: Drug: Eutonic Treprostinil Solution

INTERVENTIONS:
Drug: HypotonicTreprostinil Solution — Hypotonic Treprostinil Solution
  Other Names: Hypotonic Remodulin Solution
  Arms: Hypotonic Treprostinil Solution
Drug: Eutonic Treprostinil Solution — Eutonic Treprostinil Solution
  Other Names: Eutonic Remodulin Solution
  Arms: Eutonic Treprostinil Solution

SUMMARY:
The investigators will test whether hypotonic (diluted) remodulin solution causes less pain than the eutonic (undiluted) solution supplied by the manufacturer.

ELIGIBILITY:
Inclusion Criteria:

* PAH by standard criteria
* Treatment with subcutaneous remodulin infusion for at least 3 months, with stable dose for 1 month
* Pain at infusion site (defined as > 8 on McGill Pain Questionnaire)

Exclusion Criteria:

* Known pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Daily Pain Diary | 2 weeks

SECONDARY OUTCOMES:
McGill Pain Questionnaire | 2 weeks
CAMPHOR quality of life questionnaire | 2 weeks
6 minute walk distance | 2 weeks
NT-proBNP level | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Langleben, MD, Study Chair — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada